CLINICAL TRIAL: NCT02825654
Title: CSP #595 - Pulmonary Health and Deployment to Southwest Asia and Afghanistan
Brief Title: Service and Health Among Deployed Veterans
Acronym: SHADE
Status: Enrolling by invitation | Type: Observational
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: United States Department of Defense (U.S. Federal Agency); Harvard University (Other)
Responsible Party: Sponsor
Other Study IDs: 595
Record Dates: First submitted 2016-06-21; First posted 2016-07-07 (Estimated); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Pulmonary Function
Keywords: Pulmonary; Lung; Military and environmental exposures; Epidemiologic; Observational; Interview or questionnaire; Deployment related; Enduring Freedom; Iraqi Freedom

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 50 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Post-9/11 Gulf War Era Veterans: Military personnel who deployed to Central Asia, Southwest Asia, and Africa during the Post-9/11 Gulf War Era

SUMMARY:
The purpose of the study is to better understand the health, including lung health, of Veterans who deployed in support of Operation Enduring Freedom (OEF), Operation Iraqi Freedom (OIF), or Operation New Dawn (OND) and other deployments following these Operations.

DETAILED DESCRIPTION:
The aim of the study is to characterize the impact of deployment-related pollution exposures during the Post-9/11 Gulf War Era on current respiratory health using objectively ascertained and standardized physiologic and epidemiologic measures. The primary objective in support of this aim is to assess the association of cumulative exposure to PM2.5 during deployments to the U.S. bases and other locations in Central Asia (Afghanistan and Kyrgyzstan), Southwest Asia (Iraq, Kuwait, Qatar, and United Arab Emirates) and Africa (Djibouti) with current measures of pulmonary function. Secondary objectives in support of the aim will examine the association of cumulative exposure to PM2.5 during deployments with the clinical outcome of medically-treated asthma. The investigators will also explore the impact of deployment duration on both pulmonary function and asthma.

This study will execute 4 distinct efforts to meet the study objectives: (1) enroll a study cohort of up to 6,200 Veterans who live within the catchment area of 6 VA recruitment sites, conduct an in-person assessment of pulmonary function, and collect data on key covariates; (2) create a spatial-temporal exposure grid of environmental PM2.5 levels averaged per week per 1 square kilometer at locations where military personnel served; (3) link each individual's location and duration (spatial-temporal) history during deployed and non-deployed times with averaged PM exposures during each of these time periods; and (4) conduct association analyses to test hypotheses of deployment-related cumulative PM2.5 exposure and current respiratory health by combining exposure data with data collected from the cohort members and from their military records.

ELIGIBILITY:
Inclusion Criteria:

* Served during the Post-9/11 Gulf War Era in a service branch that had land-based deployments (Air Force, Army, and Marine Corps)
* Deployed to Afghanistan, Kyrgyzstan, Iraq, Kuwait, Qatar, United Arab Emirates, or Djibouti between October 1, 2001 and August 31, 2021

Exclusion Criteria:

* Active duty at the time of recruitment
* Impaired decision making capacity
* No English language proficiency
* Prisoners

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The sampling frame for the study is military personnel identified from Department of Defense (DoD) Defense Manpower Data Center (DMDC) records who meet the inclusion and exclusion criteria. From among those Veterans who meet study eligibility, the investigators will identify a sample of Veterans living in the catchment area of the participating VA medical centers for recruitment. The study is not open to volunteers; Veterans must be selected from the sampling frame to participate.
Sampling Method: Probability Sample
Enrollment: 6200 (Estimated)
Dates: Start 2018-03-08 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Current forced expiratory volume in 1 second (FEV1) | Outcome measured at time of in-person study visit (Day 1)
  An assessment of pulmonary function obtained through spirometry

SECONDARY OUTCOMES:
Current forced vital capacity (FVC) | Outcome measured at time of in-person study visit (Day 1)
  An assessment of pulmonary function obtained through spirometry
Current FEV1/FVC ratio | Outcome measured at time of in-person study visit (Day 1)
  An assessment of pulmonary function obtained through spirometry
Pharmaceutically-treated asthma | Outcome measured at time of in-person study visit (Day 1)
  Based on medication inventory, the investigators will classify medically-treated asthma therapy into mild, moderate, and severe based on the intensity of asthma therapy as suggested by the Global Strategy for Asthma Management and Prevention, Global Initiative for Asthma (GINA) 2015.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Garshick, MD, Study Chair — VA Boston Healthcare System West Roxbury Campus, West Roxbury, MA; Paul D Blanc, MD MSPH, Study Chair — San Francisco VA Medical Center, San Francisco, CA
Locations (6):
- United States (6):
  - VA San Diego Healthcare System, San Diego, CA, San Diego, California
  - Atlanta VA Medical and Rehab Center, Decatur, GA, Decatur, Georgia
  - VA Boston Healthcare System West Roxbury Campus, West Roxbury, MA, West Roxbury, Massachusetts
  - Minneapolis VA Health Care System, Minneapolis, MN, Minneapolis, Minnesota
  - Michael E. DeBakey VA Medical Center, Houston, TX, Houston, Texas
  - VA Puget Sound Health Care System Seattle Division, Seattle, WA, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
All collected data may be shared dependent upon data safeguards and IRB approvals.
Supporting Information: ICF
Time Frame: Data will be made available for sharing 1 year after the publication of the last manuscript addressing the primary aims of the study.
Access Criteria: The VA Cooperative Studies Program (CSP) has a program for sharing CSP study data: Integrated Veteran Epidemiologic Study Data Resource (INVESTD-R). The INVESTD-R website is where information is provided on CSP studies with data that can be shared for secondary analyses or to support new data collection from study members who consented to be recontacted. Data will be shared with qualifying investigators at bona fide research institutions.
URL: https://www.vacsp.research.va.gov/CSPEC/Studies/INVESTD-R/Main.asp

REFERENCES:
- [Background] Garshick E, Redlich CA, Korpak A, Timmons AK, Smith NL, Nakayama K, Baird CP, Ciminera P, Kheradmand F, Fan VS, Hart JE, Koutrakis P, Kuschner W, Ioachimescu O, Jerrett M, Montgrain PR, Proctor SP, Wan ES, Wendt CH, Wongtrakool C, Blanc PD. Chronic respiratory symptoms following deployment-related occupational and environmental exposures among US veterans. Occup Environ Med. 2024 Feb 2;81(2):59-65. doi: 10.1136/oemed-2023-109146. PMID 37968126
- [Background] Maccarone JR, Sterns OR, Timmons A, Korpak AM, Smith NL, Nakayama KS, Baird CP, Ciminera P, Kheradmand F, Fan VS, Hart JE, Koutrakis P, Jerrett M, Kuschner WG, Ioachimescu OC, Montgrain PR, Proctor SP, Redlich CA, Wendt CH, Blanc PD, Garshick E, Wan ES. Deployment-related Cigarette Smoking Behaviors and Pulmonary Function Among U.S. Veterans. Mil Med. 2024 Aug 30;189(9-10):2030-2038. doi: 10.1093/milmed/usae049. PMID 38536226
- [Background] Maccarone J, Redlich CA, Timmons A, Korpak AM, Smith NL, Nakayama KS, Baird CP, Ciminera P, Kheradmand F, Fan VS, Hart JE, Koutrakis P, Kuschner WG, Ioachimescu OC, Jerrett M, Montgrain PR, Proctor SP, Wendt CH, Wongtrakool C, Wan ES, Blanc PD, Garshick E. Sinusitis and rhinitis among US veterans deployed to Southwest Asia and Afghanistan after September 11, 2001. J Allergy Clin Immunol Glob. 2024 Oct 31;4(1):100367. doi: 10.1016/j.jacig.2024.100367. eCollection 2025 Feb. PMID 39659739
- [Background] Hosseini R, Garshick E, Slade MD, Timmons A, Korpak AM, Smith NL, Nakayama KS, Baird CP, Ciminera P, Kheradmand F, Fan VS, Hart JE, Koutrakis P, Kuschner WG, Ioachimescu OC, Jerrett M, Montgrain PR, Proctor SP, Wendt CH, Wongtrakool C, Wan ES, Blanc PD, Redlich CA. Military Inhalational Exposures Outside the Theater of Conflict and Chronic Respiratory Symptoms. JAMA Netw Open. 2025 Jul 1;8(7):e2522080. doi: 10.1001/jamanetworkopen.2025.22080. PMID 40690216
- See also: Seattle Epidemiologic Research and Information Center — http://www.seattle.eric.research.va.gov/
- See also: VA Cooperative Studies Program — http://www.research.va.gov/programs/csp/